CLINICAL TRIAL: NCT00279903
Title: Intra-articular Botulinum Toxin Type-A in Knee Osteoarthritis - a Randomized, Cortisone Controlled, Double Blind Study.
Brief Title: Is Botox Effective in Relieving Pain From Knee Osteoarthritis?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1565-05
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Botulinum Toxins, Type A; Cortisone; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cortisone (Active Comparator)
  Interventions: Drug: Cortisone
- Low Dose Btx-A (Experimental)
  Interventions: Drug: Botulinum toxin type A (Btx-A)
- High Dose Btx-A (Experimental)
  Interventions: Drug: Botulinum toxin type A (Btx-A)

INTERVENTIONS:
Drug: Botulinum toxin type A (Btx-A) — Participants randomized to Btx-A will be given either a low dose of 100 units or a high dose of 200 units. The Btx-A dose (100U or 200U) will be resonstituted with 4 cc of sterile non-preserved 0.9% sodium chloride solution.
  Other Names: Botox
  Arms: High Dose Btx-A; Low Dose Btx-A
Drug: Cortisone — 1 cc of 40 mg/cc methylprednisolone will be drawn up in 22 gauge needles with 3 cc of sterile non-preserved 0.9% sodium chloride solution.
  Other Names: Medrol
  Arms: Cortisone

SUMMARY:
Patients with painful knee osteoarthritis will be randomly allocated to one of three groups. Each group will receive a knee injection of: 1) cortisone, 2) low dose Botox, or 3) high dose Botox. Patients will then be followed for 6 months to see if they have significant pain relief or improvement in their activity level after the injection.

DETAILED DESCRIPTION:
Abstract Botulinum toxin type A (Btx-A) has been extensively studied and used clinically for its muscle paralyzing effects, but there is a growing body of evidence to support a role in pain modulation. Symptomatic osteoarthritis is a leading cause of pain, functional impairment, and disability, with significant indirect costs to society. Preliminary evidence suggests that Btx-A has a significant nociceptive effect, when injected intra-articularly, in to painful joints. The proposed study will evaluate the efficacy and safety of Btx-A injected intra-articularly in 60 subjects with moderate pain and functional impairment secondary to knee osteoarthritis, in a randomized, cortisone-controlled, double blind study, over a 6 month follow up period. If Btx-A is shown to be of equal or greater efficacy than cortisone in this patient population, it may be an excellent second line treatment for osteoarthritis, in multiple joints, where surgery is contraindicated or deferred due to age, comorbidities, or patient preference. Further studies examining the mechanism of action at the biochemical level, the clinical effect of Btx-A in other joints (in both osteoarthritis and inflammatory arthritis), the efficacy of Btx-A compared to hyaluronic acid (the only currently available injectable alternative to cortisone), and the side effect profile (effect on adjacent muscle strength, joint position sense, and long-term outcomes) would be indicated.

ELIGIBILITY:
Inclusion criteria:

1. A history of knee joint pain for greater than 6 months.
2. Medial or lateral tibiofemoral joint line tenderness.
3. Unilateral knee pain 6/10 or greater, on average, on the visual analog scale (VAS), that interferes with function most days per week.
4. Prior failed treatment with acetaminophen and/or non steroidal anti-inflammatory medications, and physical therapy (quadriceps strengthening).
5. Kellgren grade II or III radiographic changes of osteoarthritis.

Exclusion criteria:

1. Age less than 40 years.
2. Anticoagulation with warfarin or heparin.
3. Known allergy or sensitivity to any of the components of the study medications.
4. Body mass index greater than 35.
5. Previous major reconstructive surgery on the affected knee.
6. Previous arthroscopic surgery on the affected knee in the past 12 months.
7. History of crystal induced arthropathy.
8. Use of aminoglycoside antibiotics, curare-like agents, or history of neuromuscular disease such as myasthenia gravis, amyotrophic lateral sclerosis, or myopathy.
9. History of or evidence of active rheumatologic disease, diabetes, severe peripheral neuropathy, clinically evident cardiac or respiratory disease that interferes with functional status, or other serious diseases, including psychiatric disorders.
10. Evidence of recent alcohol or drug abuse, or history of medication misuse or addiction.
11. Females who are pregnant, breastfeeding, or planning a pregnancy during the study, or who think that they may be pregnant at the start of the study, or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study.
12. Intra-articular (knee) or systemic steroids in the past 6 months, or intra-articular knee hyaluronic acid injection in the past 6 months.
13. Patients who rate their average daily pain as less than 6 on a 10 point VAS scale at the screening visit.
14. Concurrent participation in another investigational drug or device study or participation in the 30 days immediately prior to study enrollment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Decrease in pain at 8 weeks post injection

SECONDARY OUTCOMES:
Improvement in function at 2, 4, 8, 12, 26 weeks
Improvement in quality of life at 2, 4, 8, 12, 26 weeks
Decrease in pain at 2, 4, 12, 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrea J. Boon, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States